CLINICAL TRIAL: NCT02951364
Title: A Post-Marketing Surveillance Study to Evaluate the Safety and Effectiveness of Harvoni Treatment Regimen in Patients With Chronic Hepatitis C Virus (HCV) Infection in Korea
Brief Title: Harvoni in Patients With Chronic Hepatitis C Virus (HCV) Infection in Korea
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-337-1966
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Hepatitis C Virus
Keywords: observational
MeSH Terms: conditions — Hepatitis C | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LDV/SOF: Adult Korean participants and pediatric Korean participants aged 12 to <18 years with genotype 1, 2, 4, 5, and 6 chronic HCV infection who are initiating commercial Harvoni regimen
  Interventions: Drug: LDV/SOF

INTERVENTIONS:
Drug: LDV/SOF — 90/400 mg tablet administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977

SUMMARY:
The primary objective of this post-marketing surveillance study is to collect and assess data related to the safety and effectiveness of Harvoni® (ledipasvir/sofosbuvir (LDV/SOF)) treatment regimen, per the approved Korea prescribing information for Harvoni, in routine clinical practice in Korea and to report the results to the Ministry of Food and Drug Safety (MFDS). Participants will be treated as part of routine practice at Korean healthcare centers by accredited physicians.

ELIGIBILITY:
Key Inclusion Criteria:

* Individuals aged 12 years and older who are living in Korea
* Adult individuals who have been informed of all pertinent aspects of the study and have voluntarily signed a Personal Information Protection Act (PIPA) consent form; Pediatric individuals who have the individuals' legally authorized representatives sign the PIPA consent form

Key Exclusion Criteria:

* Individuals treated with Harvoni outside of the approved prescribing information in Korea
* Individuals who have a contra-indication to Harvoni
* Individuals who have a contra-indication to ribavirin
* Pregnant or breastfeeding women
* Individuals who have previously been administered Harvoni
* Individuals participating in a concurrent HCV clinical trial
* Individuals planning on leaving the country during the study period

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult Korean individuals and pediatric Korean individuals aged 12 to <18 years with genotype 1, 2, 4, 5, and 6 chronic HCV infection who are initiating commercial Harvoni regimen
Sampling Method: Non-Probability Sample
Enrollment: 1081 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) and Special Situation Reports (SSRs) | Up to 30 days following treatment
  Incidence of adverse events (AEs) and special situation reports (SSRs) occurring during administration of Harvoni regimen or up to 30 days of treatments will be analyzed.
Proportion of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12) | Posttreatment Week 12
  The sustained virologic response (SVR) rate will be assessed at 12 weeks after completion (or discontinuation) of Harvoni treatment, defined as the proportion of participants with HCV RNA < lower limit of quantification (LLOQ) from 2 weeks before Posttreatment Week 12 through Posttreatment Week 24 (based on when the participant's actual visit occurs). The treatment will be assessed as "improved/success" when HCV RNA < LLOQ is achieved from 2 weeks before Posttreatment Week 12 through Posttreatment Week 24.

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) and Special Situation Reports (SSRs) | Up to Posttreatment Week 12
  Incidence of adverse events (AEs) and special situation reports (SSRs) occurring within 12 weeks after completion (or discontinuation) of treatments will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (71):
- South Korea (71):
  - CHA Bundang Medical Center, Seongnam-si, Gyeonggido
  - Hallym University Sacred Heart Hospital, Anyang-si
  - SoonChunHyang University Bucheon Hospital, Bucheon-si
  - The Catholic University of Korea Bucheon ST. Mary's Hospital, Bucheon-si
  - Bumin Hospital Haeundae, Busan
  - Inje University Haeundae Paik Hospital, Busan
  - Good Gang-An Hospital, Busan
  - Dong-A University Medical Center, Busan
  - Pusan National University Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Inje University Busan Paik Hospital, Busan
  - Busan St. Mary's Hospital, Busan
  - Busan Veterans Hospital, Busan
  - Maryknoll Medical Center, Busan
  - Changwon Fatima Hospital, Changwon
  - Dankook University Hospital, Cheonan
  - SoonChunHyang University Cheonan Hospital, Cheonan
  - Hallym University ChunCheon Sacred Heart Hospital, Chuncheon
  - Konkuk University Chungju Hospital, Chungju
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Medical Center, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Kyungpook national university medical center Chil-Gok, Daegu
  - Chungnam National University Hospital, Daejeon
  - Konyang University Hospital, Daejeon
  - GangNeung Asan Hospital, Gangneung-si
  - Dongguk University Ilsan Hospital, Goyang
  - Myongji Hospital, Goyang
  - National Health Insurance Corporation Ilsan Hospital, Goyang-si
  - Kumi Cha Hospital, Gumi
  - Chosun University Hospital, Gwangju
  - Kwangju Christian Hospital, Gwangju
  - Hanyang University Guri Hospital, Gyeonggi-do
  - Dongguk University Gyeongju Hospital, Gyeongju
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si
  - Chonnam National University Hwasun Hospital, Hwasun
  - WonKwang University Hospital, Iksan
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Incheon
  - Inha University Hospital, Incheon
  - Gachon University Gil Medical Center, Incheon
  - Cheju Halla General Hospital, Jeju City
  - Presbyterian Medical Center, Jeonju
  - Chonbuk National University Hospital, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Seoul National University Bundang Hospital, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Seoul
  - SoonChunHyang University Hospital, Seoul
  - Hanyang University Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - SMG - SNU Boramae Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Inje University Seoul Paik Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Eulji General Hospital, Seoul
  - Inje University Sanggye Paik Hospital, Seoul
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon
  - The Catholic University of Korea Uijeongbu St. Mary's Hospital, Uijeongbu-si
  - Ulsan University Hospital, Ulsan
  - DongKang Hospital, Ulsan
  - Ulsan Hospital, Ulsan
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No